CLINICAL TRIAL: NCT06586359
Title: Evaluation of Bone Mineral Density in Patients with Childhood-onset Systemic Lupus Erythematous, in Relation to Disease Clinical Criteria
Brief Title: Bone Mineral Density in Patients with Childhood-onset Systemic Lupus Erythematous, in Relation to Disease Clinical Criteria
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Shehata Abdelmohsen Issa, 71515,Assiut, Assiut University
Other Study IDs: childhood-onset systemic lupus
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erthematosus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
* To determine the most common clinical characteristics in patients with childhood -onset systemic lupus erythematosus.
* To detect prevalence of low bone mineral density in patients with childhood -onset systemic lupus erythematosus.

DETAILED DESCRIPTION:
Childhood-onset systemic lupus erythematosus (CSLE) is a chronic, inflammatory, autoimmune disease that is characterized by multisystemic involvement with diverse clinical presentation and can involve one or more organ (1).This condition has a broad spectrum of clinical features ranging from mild cutaneous involvement to severe organ damage, such as kidney failure, pulmonary hypertension, and cardiac failure. The diagnosis of SLE is based on clinical and laboratory findings (2).The disease has a variable prevalence across the globe, with higher prevalence in low to middle income Asian and African countries than previously thought (3,4). Despite being common in young age females of reproductive age, the pediatric populations also suffer from lupus, where it has more aggressive disease course and complications (5).

Over the years, the management of CSLE has improved significantly, increasing the life expectancy of affected individuals however, CSLE patients still face numerous challenges, such as the increased risk of developing secondary complications like osteoporosis(6).

Osteoporosis, a skeletal disorder characterized by compromised bone strength and an increased risk of fractures, is a major public health concern worldwide (7). The association between CSLE and osteoporosis has been studied extensively and there is evidence suggesting an increased risk of osteoporosis in patients with CSLE (8) ,Possible factors contributing to low bone mineral density in CSLE patients include chronic inflammation, glucocorticoid therapy, and the presence of various cytokines produced by immune cells that interfere with bone homeostasis. Lifestyle factors and low vitamin D levels in CSLE patients may further contribute to the risk of osteoporosis (9,10).

Among children and adolescents, the recommended technology for clinical measurement of bone mineral density (BMD) and bone mineral content (BMC) is dual energy X-ray absorptiometry (DXA). It is a radiological method that detects the attenuation of two photon beams of different energies as they pass through the soft tissue and bone. DXA remains a method of choice because of its availability, low ionising radiation exposure, precision, scan speed(11). Mostly, the posteroanterior lumbar spine (L1-L4) and the total body less head (TBLH) are the skeletal sites of choice. Other sites such as the proximal femur, distal radius and lateral distal femur can be used to measure BMD if assessing standard sites are not feasible, and appropriate reference DXA data are available (12).

In recent years, studies have shown that vitamin D deficiency in patients with CSLE is strongly associated with reduced bone mineral density (BMD) determined by (DXA)(13).Vitamin D inadequacy is highly prevalent in CSLE patients due to the avoidance of sunshine, photoprotection, renal insufciency and the use of medications such as glucocorticoids, anticonvulsants, antimalarials and the calcineurin inhibitors, which alter the metabolism of vitamin D or down regulate the functions of the vitamin D receptor (14).

This study aims to disscus the clinical criteria in patients diagnosed as CSLE at Assiut University Children's Hospital ,and to asses bone mineral density based on (DXA) and 25(OH) vitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients below 18 years old.
2. Both sexes.
3. The Patients should be diagnosed as SLE, according to 2019 European league against rheumatism (EULAR)/ American college of rheumatology (ACR) SLE classiﬁcation criteria from >6 months ago.

Exclusion Criteria:

1. Patients with autoimmune diseases other than CSLE.
2. Patients not fulfilling the criteria for diagnosis of CSLE.
3. Active infections.
4. Malignancies.
5. Patients with other diseases which decrease vitamin D levels as malabsorption, cholestatic jaundice and chronic kidney disease.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Patients diagnosed as SLE, according to 2019 European league against rheumatism (EULAR)/ American college of rheumatology (ACR) SLE classiﬁcation criteria from >6 months ago.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Detection of prevalence of low bone mineral density and clinical characteristics in patients with childhood -onset systemic lupus erythematosus | Baseline
  There is association between SlE and bone mineral density. Possible factors contributing to low bone mineral density in CSLE patients include chronic inflammation, glucocorticoid therapy, and the presence of various cytokines produced by immune cells that interfere with bone homeostasis. Lifestyle factors and low vitamin D levels in CSLE patients may further contribute to the risk of osteoporosis

REFERENCES:
- [Background] Kiriakidou M, Ching CL. Systemic Lupus Erythematosus. Ann Intern Med. 2020 Jun 2;172(11):ITC81-ITC96. doi: 10.7326/AITC202006020. PMID 32479157
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus. Arthritis Rheumatol. 2019 Sep;71(9):1400-1412. doi: 10.1002/art.40930. Epub 2019 Aug 6. PMID 31385462
- [Background] Tian J, Zhang D, Yao X, Huang Y, Lu Q. Global epidemiology of systemic lupus erythematosus: a comprehensive systematic analysis and modelling study. Ann Rheum Dis. 2023 Mar;82(3):351-356. doi: 10.1136/ard-2022-223035. Epub 2022 Oct 14. PMID 36241363